CLINICAL TRIAL: NCT04190446
Title: A Randomized, Parallel Phase II Trial of Hypofractionated Proton Therapy or IMRT for Recurrent, Oligometastatic Prostate Cancer Involving Only Pelvic and/or Para-Aortic Lymph Nodes Following Primary Localized Treatment
Brief Title: A Study to Evaluate Hypofractionated Proton Therapy or IMRT for Recurrent, Oligometastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1851; NCI-2019-07705 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1851 (Other: Mayo Clinic in Rochester); 19-000708 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Prostate Adenocarcinoma; Oligometastatic Prostate Carcinoma; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Proton Therapy; Protons; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (proton beam radiation therapy) (Experimental): Patients undergo proton beam radiation therapy 5 days a week over 3 weeks. Patients undergo PET scan, CT scan, MRI, and blood sample collection throughout the study.
  Interventions: Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection
- Arm II (IMRT) (Experimental): Patients undergo IMRT 5 days a week over 5 weeks. Patients undergo PET scan, CT scan, MRI, and blood sample collection throughout the study.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Questionnaire Administration; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm II (IMRT)
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; Radiation, Proton Beam; External beam radiation therapy protons (procedure); emission tomography (procedure); positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Arm I (proton beam radiation therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm I (proton beam radiation therapy)
Other: Questionnaire Administration — Ancillary studies
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging; Structural MRI; sMRI
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II trial studies the side effects of radiation therapy (hypofractionated proton beam therapy or IMRT) for the treatment of prostate cancer that has come back (recurrent) or that has spread to a limited number of sites (oligometastatic) following primary localized treatment. Hypofractionated proton beam radiation therapy delivers smaller doses of radiation therapy over time and may kill more tumor cells and have fewer side effects. IMRT uses high energy x-rays to kill tumor cells and shrink tumors. This trial is being done to find out if a shorter course of radiation therapy is better with fewer side effects for patients with recurrent prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess late >= grade 3 gastrointestinal (GI) and/or genitourinary (GU) toxicity of interest with the hypofractionated regimen with proton beam therapy or intensity-modulated radiation therapy (IMRT) (late defined as 3 to 24 months after protocol radiation therapy [RT]).

SECONDARY OBJECTIVES:

I. Late grade >= 2 GI and/or GU toxicities of interest within 24 months after the protocol RT, using the Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.0.

II. Acute grade >= 3 GI and/or GU toxicities of interest during and within 3 months after the protocol RT, using the CTCAE v4.0.

III. Compare the rates of late >= grade 3 GI and/or GU toxicity between the 2 treatment schedules.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo proton beam radiation therapy 5 days a week over 3 weeks. Patients undergo positron emission tomography (PET) scan, computed tomography (CT) scan, magnetic resonance imaging (MRI), and blood sample collection throughout the study.

ARM II: Patients undergo IMRT 5 days a week over 5 weeks. Patients undergo PET scan, CT scan, MRI, and blood sample collection throughout the study.

After completion of study, patients are followed up at 3-6, 12, 18, 24, 30, 36, 42, 48, 54, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Male; age >= 18 years
* Histological confirmation of prostate adenocarcinoma
* Recurrent prostate cancer after prior receipt of primary radiotherapy to the prostate (can also include treatment of splenic vessels [SVs] and lymph nodes [LNs]) or salvage RT to the prostate fossa (can also include prior pelvic RT)
* Oligometastatic extent of disease

  * Recurrent disease involving lymph nodes as diagnosed with choline positron emission tomography (PET)/computed tomography (CT) or other advanced PET imaging (prostate-specific membrane antigen [PSMA] or flucyclovine)
  * Limited to pelvic and/or retroperitoneal/para-aortic lymph nodes
* Zubrod performance score (PS) =< 1
* Signed informed consent

Exclusion Criteria:

* Bone or visceral metastases present
* Lymph node metastases beyond the pelvis and/or retroperitoneum
* Contraindications to RT (e.g., uncontrolled inflammatory bowel disease)
* Contraindications to androgen suppression
* Concurrent antineoplastic agents (chemotherapy)
* Previous or concurrent malignancy other than non-melanoma skin cancer within 5 years of diagnosis of prostate cancer
* Inability to start the radiation portion of the protocol treatment within 6 months after study enrollment
* Medical or psychiatric conditions that preclude informed decision-making or compliance with the protocol treatment or follow-up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2028-11-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of late > grade 3 GI and/or GU toxicity | Up to 24 months after RT
  Assessed by the number of patients who experience a late (≥ 90 days after RT start date) grade 3 or higher gastrointestinal (GI) and/or genitourinary (GU) adverse event (AE) defined as possibly, probably, or definitely related to radiation therapy (RT). Adverse events will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Incidence of acute adverse events | Up to 3 months after the completion of RT
  Assessed by the number of patients with >= grade 3 GI or GU acute adverse events. Acute AEs are defined as those that occur from day 1, or commencement of RT, through 3 months after the completion of protocol treatment.
Incidence of late adverse events | Between 3 months and 2 years after completion of proton beam therapy
  Assessed by the number of ≥ grade 2 GI or GU late adverse events per CTCAE v 4.0 will be recorded. A late AE is defined as an adverse event that occurs any time between 3 months and 2 years after completion of proton beam therapy.
Incidence of grade 3 or higher GI or GU adverse events per treatment schedule | Up to 60 months
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Rates of late ≥ grade 3 GI and/or GU toxicity will be compared between the treatment schedules.
Incidence of adverse events Incidence of adverse events Incidence of adverse events | Up to 60 months
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient.

OTHER OUTCOMES:
Expanded Prostate Cancer Index Composite short form (EPIC-26) questionnaire | Baseline, up to 60 months
  The EPIC-26 questionnaire is a 26-item questionnaire used to assess health-related quality of life (HRQOL). Items are scores on a Likert-type scales such as 0-4 where 0=no problem and 4=big problem. Higher scores indicate better HRQOL.
Disease-free survival | Up to 60 months
  Defined as the time from registration until the time of the first occurrence of biochemical failure, local recurrence, regional recurrence, distant metastases, or death due to any cause
Disease-specific survival | Up to 60 months
  Defined as the time from registration until death due to prostate cancer (death attributed to carcinoma of the prostate by the investigator or death due to complications of treatment)
Overall survival | Up to 60 months
  Defined as the time from registration until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Davis, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials